CLINICAL TRIAL: NCT02197195
Title: The Role of Chocolate Milk and Fruit Drink on Subjective Appetite and Glycaemic Response With or Without Exercise in Normal Weight 9-14 Year Old Boys
Brief Title: Sugars-sweetened Beverages and Exercise on Glycaemic Response and Subjective Appetite in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assistant Professor, School of Nutrition, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2013-251
Record Dates: First submitted 2014-07-20; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Glycemic Control; Subjective Appetite
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chocolate Milk Beverage (Experimental): Chocolate milk beverage and sitting quietly
  Interventions: Dietary Supplement: Chocolate Milk
- Chocolate Milk Beverage and Exercise (Experimental): Chocolate milk beverage and exercising
  Interventions: Dietary Supplement: Chocolate Milk; Behavioral: Exercise
- Fruit Drink Beverage (Experimental): Fruit drink beverage and sitting quietly
  Interventions: Dietary Supplement: Fruit Drink
- Fruit Drink Beverage and Exercise (Experimental): Fruit drink beverage and exercising
  Interventions: Dietary Supplement: Fruit Drink; Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: Chocolate Milk
  Arms: Chocolate Milk Beverage; Chocolate Milk Beverage and Exercise
Dietary Supplement: Fruit Drink
  Arms: Fruit Drink Beverage; Fruit Drink Beverage and Exercise
Behavioral: Exercise
  Arms: Chocolate Milk Beverage and Exercise; Fruit Drink Beverage and Exercise

SUMMARY:
The purpose of the study is to understand the role chocolate milk compared to a fruit drink, with and without exercise, on glycaemic regulation and subjective appetite in children. The investigators hypothesize that chocolate milk in combination with exercise will have the greatest effect attenuating glycaemic response. Blood glucose will be measured by finger prick following drink consumption (0 min) and exercise or sitting (15 min), and at 65 minutes. Subjective appetite will be measured at 0, 20, 35, 50 and 65 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, boy, born at full term and normal birth weight

Exclusion Criteria:

* Girls, have significant learning, behavioral, or emotional difficulties

Ages: 9 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Blood Glucose (mmol/L) | at baseline (0), 20 and 65 minutes
  Blood Glucose (mmol/L) determined by fingerprick glucometer reading

SECONDARY OUTCOMES:
Subjective Appetite (mm) | 0 - 65 mins
  Subjective appetite (in mm) determined by visual analogue scale will be determined at 0, 20, 35, 50 and 65 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryerson University, Toronto, Ontario, Canada